CLINICAL TRIAL: NCT00809003
Title: Assessment of Inflammatory and Functional Changes in the Ocular Surface Associated With Dry Eye Disease
Acronym: JADE
Status: Completed | Type: Observational
Sponsor: University of Waterloo (Other)
Collaborators: Alcon Research (Industry)
Responsible Party: Dr Craig Woods, CCLR
Other Study IDs: P/269/07/L
Record Dates: First submitted 2008-12-12; First posted 2008-12-16 (Estimated); Last update posted 2008-12-16 (Estimated); Status verified 2008-12

CONDITIONS: Sjogren's Syndrome; Dry Eye
Keywords: Non dry eyed(normals)
MeSH Terms: conditions — Sjogren's Syndrome; Dry Eye Syndromes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Sjogren's group
- Dry eye
- Normals

SUMMARY:
This project will examine the similarities and differences of the ocular surface and tear film in patients with Sjogren's syndrome related to dry eye, severe dry eye and those who do not have dry eye. This knowledge will help clinicians understand the processes that create these dry eye conditions and will strengthen the treatment and management strategies that will be used. The subjects will participate in a series of dry eye tests that they have already experienced in clinic, along with the gathering of tear samples and surface cells. These tissues will then be analyzed at a distant site.

DETAILED DESCRIPTION:
Dry eye is a multifactorial disease of the tears and ocular surface that results in symptoms of discomfort, visual disturbance and tear film instability with potential damage to the ocular surface. It is accompanied by increased osmolarity of the tear film and inflammation of the ocular surface. A number of factors have been implicated in triggering this disease, including age, hormone changes and autoimmune disease.

Sjogren's syndrome(SS) is a common autoimmune disorder, characterized by chronic inflammatory infiltration of exocrine glands (particularly salivary and lacrimal) and systemic immune reactivity, resulting in dry eye and dry mouth. The mechanism of inflammation of the lacrimal gland in these patients is well documented. It is believed that these pathological changes facilitate the secretion of inflammatory biochemicals on to the ocular surface. Additionally, in SS, there are also pathological changes to epithelial cells of the cornea and conjunctiva (such as upregulation of mRNAs coding for inflammatory cytokines) which subsequently contribute to the increased secretion of the cytokines themselves. Taken together, these changes result in an increased concentration of inflammatory mediators in the tear film, which then drive the propagation of the dry eye disease process. Severe dry eye (DE) patients present with a very similar clinical outcome to SS patients, however, inflammatory processes associated with either the initiation or propagation of their dry eye disease has not been well characterized.

This research project was established to quantify similarities and / or differences between SS and severe dry eye participants, with respect to ocular surface inflammation and function. Specifically, this study will examine dry eye symptoms, ocular surface integrity and tear film volume and flow. Additionally, the concentration of inflammatory cytokines present in the tear film will be quantified.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria (Sjogren's group)

A person is eligible for inclusion in the study, for the dry eye group, if she:

1. Has been diagnosed to have SS(confirmed via American-European Consensus Criteria 2002)and dry eye and half of the time wants to use eye drops for dry eye symptoms (dry eye group).
2. Has read, understood and signed an information consent letter.
3. Is willing and able to follow instructions and maintain the appointment schedule.
4. Has had an ocular examination in the last two years.

Inclusion criteria (severe DE group)

A person is eligible for inclusion in the study, for the dry eye group, if he/she:

1. Has moderate or severe dry eye symptoms based on dry eye questionnaire and half of the time wants to use eye drops for dry eye symptoms (dry eye group)
2. Has read, understood and signed an information consent letter.
3. Is willing and able to follow instructions and maintain the appointment schedule.
4. Has had an ocular examination in the last two years.

Inclusion criteria (control group)

A person is eligible for inclusion in the study, for the control group, if he/she:

1. Has read, understood and signed an information consent letter.
2. Is willing and able to follow instructions and maintain the appointment schedule.
3. Has clear corneas and no active ocular disease.
4. Has had an ocular examination in the last two years.

Exclusion Criteria:

A person will be excluded from the study if he/she (Sjogren's group):

1. Is a contact lens wearer.
2. Has any clinically significant belpharitis.
3. Has undergone corneal refractive surgery.
4. Is aphakic.
5. Has any active ocular disease.
6. Is using any systemic or topical medications that may affect ocular health.
7. Has known sensitivity to the diagnostic pharmaceuticals to be used in the study.
8. Is participating in any other type of clinical or research study.

A person will be excluded from the study if he/she (Dry eye group):

1. Is a contact lens wearer.
2. Has any clinically significant belpharitis.
3. Has undergone corneal refractive surgery.
4. Is aphakic.
5. Has any active ocular disease.
6. Is using any systemic or topical medications that may affect ocular health.
7. Has known sensitivity to the diagnostic pharmaceuticals to be used in the study.
8. Is participating in any other type of clinical or research study.

A person will be excluded from the study if he/she (control group):

1. Has rheumatoid arthritis, diabetes, Sjogren's syndrome or any other systemic disease affecting ocular health.
2. Is using any systemic or topical medications (other than eye drops for dry eye symptoms) that may affect ocular health and neuro-endocrine system function.
3. Has undergone corneal refractive surgery.
4. Is aphakic.
5. Has any active ocular disease.
6. Has known sensitivity to the diagnostic pharmaceuticals to be used in the study.
7. Is participating in any other type of clinical or research study.
8. Is a contact lens wearer.
9. Has blepharitis.

Ages: 17 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Primary care
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2007-09; Study Completion 2007-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Desmond Fonn, MOptom, Principal Investigator — University of Waterloo
Locations (1):
- Centre for Contact Lens Research, School of Optometry, Waterloo, Ontario, Canada